CLINICAL TRIAL: NCT02054871
Title: Randomised Controlled Trial to Evaluate the Reno-protective Benefits of Remote Ischaemic Preconditioning in Patients Undergoing Infrainguinal Peripheral Angioplasty
Brief Title: RCT to Evaluate the Renal Protective Effects of Remote Ischaemic Preconditioning in Peripheral Angioplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mid Western Regional Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Stewart Walsh, Consultant Vascular Surgeon, Mid Western Regional Hospital, Ireland
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MWRH09644
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Peripheral Vascular Disease
Keywords: Peripheral Angioplasty; Remote Ischaemic Preconditioning; Contrast Induced Nephropathy
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EGFR 30-60 (Experimental): Experimental: RIPC Remote preconditioning Calculated EGFR based on MDRD. Patients receive intravenous fluids preprocedure as additional renal protection.
  Preconditioning will be performed in the same manner as several previous trials. Immediately prior to angiography a CE-approved blood pressure cuff will be placed around one arm of the patient. It will then be inflated to a pressure of 200mmHg for 5 minutes. For patients with a systolic blood pressure >185mmHg, the cuff will be inflated to at least 15mmHg above the patient's systolic blood pressure. The cuff will then be deflated and the arm allowed reperfuse for 5 minutes. This will be repeated so that each patient receives a total of 4 ischaemia-reperfusion cycles.
  Interventions: Procedure: RIPC
- EGFR 60-90 (Experimental): Experimental: RIPC Remote preconditioning. EGFR calculated using MDRD equation. Oral hydration pre-procedural as reno-protective measure. Preconditioning will be performed in the same manner as several previous trials. Immediately prior to angiography a CE-approved blood pressure cuff will be placed around one arm of the patient. It will then be inflated to a pressure of 200mmHg for 5 minutes. For patients with a systolic blood pressure >185mmHg, the cuff will be inflated to at least 15mmHg above the patient's systolic blood pressure. The cuff will then be deflated and the arm allowed reperfuse for 5 minutes. This will be repeated so that each patient receives a total of 4 ischaemia-reperfusion cycles.
  Interventions: Procedure: RIPC
- EGRF 30-60 (No Intervention): No Intervention: Remote preconditioning control Calculated EGFR based on MDRD. Patients receive intravenous fluids preprocedure as additional renal protection.
  Patients randomised to this group will receive routine care.
- EGRF 60-90 (No Intervention): No Intervention: Remote preconditioning control EGFR calculated using MDRD equation. Oral hydration pre-procedural as reno-protective measure. Patients randomised to this group will receive routine care.

INTERVENTIONS:
Procedure: RIPC — A standard, CE-approved tourniquet cuff will be placed around one arm of the patient. It will then be inflated to a pressure of 200mmHg for 5 minutes. For patients with a systolic blood pressure >185mmHg, the cuff will be inflated to at least 15mmHg above the patient's systolic blood pressure. The cuff will then be deflated and the arm allowed reperfuse for 5 minutes. This will be repeated so that each patient receives a total of 3 ischaemia-reperfusion cycles. Additional, blood and urine samples will be collected on Day 1, Day 2 and Day 3 post procedure.
  Arms: EGFR 30-60; EGFR 60-90

SUMMARY:
This study aims to demonstrate if remote ischaemic preconditioning (RIPC) may confer renal protection in patients undergoing peripheral angioplasty. Patients will be randomised to receive RIPC and biomarkers for renal injury will be analysed post procedure to determine if any protective benefit was obtained.

DETAILED DESCRIPTION:
Ischaemic preconditioning is an endogenous mammalian mechanism whereby a brief period of ischaemia and reperfusion confers resistance to subsequent prolonged ischaemic insults. First observed in the canine heart, subsequent investigators noted that brief ischaemia in remote organs e.g. skeletal muscle, induced protection in key central organs e.g. the heart. This remote ischaemic preconditioning (RIPC) does not require direct interference with the target organs' blood supply. It can be induced using blood pressure cuffs to produce brief episodes of upper limb ischaemia and reperfusion and confers protection upon numerous organs simultaneously. RIPC reduces myocardial injury following aortic aneurysm repair, cardiac surgery and angioplasty. It also reduces adverse ischaemic events up to six months following percutaneous coronary intervention, implying some medium-term effect.

To date ischaemic conditioning has been applied primarily to the heart however animal studies have shown pre conditioning to offer renal protection.

Fikret et al in 2012 in the Renal Protection Trial demonstrated a protective benefit with RIPC from the development of CIN in high risk patients undergoing elective coronary angiography.Whittaker and Przyklenk in 2011 explored this concept retrospectively using data from patients who had undergone emergency angioplasty for ST elevation myocardial infarction. The original trial was a RCT which examined the protective effect of postconditioning on myocardial ischemia. The authors retrospectively examined if study patients treated with multiple coronary balloon inflations had better renal function than patients not exposed to this remote conditioning. They concluded that patients in the conditioning group received 25% more contrast volume than the control group and showed no decline in renal function as demonstrated by examination of glomular filtration rate at day 3 post procedure in comparison to the control group which saw a significant decline in renal function. The need for contrast-based procedures is rising, with increasing numbers of patients undergoing endovascular procedures, as is the incidence of postcontrast renal failure, which has a reported mortality of 34%. The potential use of RIPC therefore to reduce the risk of kidney damage needs further investigation in a prospective study and the PAD patient group who are routinely exposed to contrast administration in angiography are an ideal study group.

ELIGIBILITY:
Inclusion Criteria:

* Elective intra-arterial, infrainguinal peripheral angiography/angioplasty
* Written informed consent
* Patients >18yrs of age
* Patients with CKD (Stage2/3) as evidenced by eGFR <90ml/min/1.73m2

Exclusion Criteria:

* Severe renal impairment eGFR <30ml/min
* Evidence of acute renal failure or patients on dialysis
* History of previous CIN
* Contraindication to intravenous volume replacement therapy
* Pregnancy
* Patients on glibenclamide or nicorandil (these medications may interfere with RIPC)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-07 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Renal impairment | 72 hours post procedural
  Serial assessment of renal biomarkers in serum and urine in 72 hour period post procedure

SECONDARY OUTCOMES:
Anti-inflammatory effect of RIPC | 3-6 months post recruitment
  Assessment of additional postulated benefits of anti-inflammatory effects with RIPC in terms of decreased restenosis rates and lower inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Walsh, MCh FRCS, Principal Investigator — University of Limerick
Locations (1):
- HSE Mid Western Regional Hospital, Limerick, Limerick, Ireland

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250